CLINICAL TRIAL: NCT02098109
Title: A Randomized, Open Label, Non-inferiority Study of XM02 Filgrastim (Granix) and Filgrastim (Neupogen) When Administered in Combination With Plerixafor for Autologous Stem Cell Mobilization in Patients With Multiple Myeloma or Non-Hodgkin Lymphoma
Brief Title: Non-inferiority Study of XM02 Filgrastim (Granix) and Filgrastim (Neupogen) in Combination With Plerixafor for Autologous Stem Cell Mobilization in Patients With Multiple Myeloma or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201403068
Record Dates: First submitted 2014-03-20; First posted 2014-03-27 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Multiple Myeloma; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim; Blood Component Removal; plerixafor; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XM02 Filgrastim (Granix) and Plerixafor (Experimental): * XM02 Filgrastim (Granix) 10 mg/kg Days 1 through 4 (Days 5 through 8 may be required if target collection goal has not be met)
  * Plerixafor 0.24 mg/kg Day 4 (Days 5 through 7 may be required if target collection goal has not be met)
  * Apheresis on Day 5 (may need to be done on Days 6-8 if target collection goal has not been met)
  * Patients who undergo infusion of the mobilized PBSC product within 6 months of the last apheresis procedure will be followed through Day +100 post-infusion (+/- 30 days) to assess for transplant outcomes (neutrophil and platelet engraftment, and readmission rate). Patients who successfully mobilize > 2.0 x 10^6 CD34+ cells/kg but do not undergo infusion of the mobilized PBSC product within 6 months of the last apheresis procedure will be discontinued from follow-up.
  Interventions: Drug: XM02 Filgrastim; Procedure: Apheresis; Drug: Plerixafor; Procedure: Stem Cell Transplant
- Filgrastim (Neupogen) and Plerixafor (Active Comparator): * Filgrastim (Neupogen) 10 mg/kg Days 1 through 4 (Days 5 through 8 may be required if target collection goal has not be met)
  * Plerixafor 0.24 mg/kg Day 4 (Days 5 through 7 may be required if target collection goal has not be met)
  * Apheresis on Day 5 (may need to be done on Days 6-8 if target collection goal has not been met)
  * Patients who undergo infusion of the mobilized PBSC product within 6 months of the last apheresis procedure will be followed through Day +100 post-infusion (+/- 30 days) to assess for transplant outcomes (neutrophil and platelet engraftment, and readmission rate). Patients who successfully mobilize > 2.0 x 10^6 CD34+ cells/kg but do not undergo infusion of the mobilized PBSC product within 6 months of the last apheresis procedure will be discontinued from follow-up.
  Interventions: Drug: Filgrastim; Procedure: Apheresis; Drug: Plerixafor; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: XM02 Filgrastim
  Other Names: Granulocyte Colony-Stimulating Factor, G-CSF, Recombinant Methionyl Human G-CSF, tbo-filgrastim, Granix
  Arms: XM02 Filgrastim (Granix) and Plerixafor
Drug: Filgrastim
  Other Names: Neulasta®, Neupogen®, Granulocyte Colony-Stimulating Factor, G-CSF
  Arms: Filgrastim (Neupogen) and Plerixafor
Procedure: Apheresis
Drug: Plerixafor
  Other Names: Mozobil, AMD3100
Procedure: Stem Cell Transplant
  Other Names: ASCT

SUMMARY:
This study will compare the results of stem cell mobilization using drugs called filgrastim (Neupogen) and plerixafor with the results of stem cell mobilization using drugs called XM02 filgrastim (Granix) and plerixafor.

DETAILED DESCRIPTION:
This study will compare the results of stem cell mobilization using drugs called filgrastim (Neupogen) and plerixafor with the results of stem cell mobilization using drugs called XM02 filgrastim (Granix) and plerixafor. The FDA has determined that Granix is biosimilar to Neupogen, which means that they are similar in terms of quality, safety, and efficacy; however, Granix has not been tested in the context of stem cell mobilization to see how its effectiveness compares to that of Neupogen

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of multiple myeloma or non-Hodgkin lymphoma
* Eligible for autologous transplantation
* Adequate bone marrow function as defined as:

  * White Blood Cell Count ≥ 3.0x109/L
  * Absolute Neutrophil Count ≥ 1.5x109/L
  * Platelet Count ≥ 100x109/L
* Able to understand and willing to sign an IRB-approved informed consent document
* Surgically or biologically sterile or willing to practice acceptable birth control, as follows:

  * Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of Day 1 of study treatment. Women of childbearing potential must agree to abstain from sexual activity or use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period. Acceptable methods of birth control include: barriers (condoms), oral contraceptive, intrauterine device (IUD), transdermal/implanted or injected contraceptives, and abstinence
  * Males must agree to abstain from sexual activity or agree to utilize a medically approved contraception method during and for 3 months after the treatment period. Acceptable methods of birth control include: barriers (condoms), oral contraceptive, intrauterine device (IUD), transdermal/implanted or injected contraceptives, and abstinence

Exclusion Criteria:

* Previous autologous stem cell collection
* Known hypersensitivity to filgrastim, plerixafor, or E. coli derived products
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Abboud, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhamidipati PK, Fiala MA, Grossman BJ, DiPersio JF, Stockerl-Goldstein K, Gao F, Uy GL, Westervelt P, Schroeder MA, Cashen AF, Abboud CN, Vij R. Results of a Prospective Randomized, Open-Label, Noninferiority Study of Tbo-Filgrastim (Granix) versus Filgrastim (Neupogen) in Combination with Plerixafor for Autologous Stem Cell Mobilization in Patients with Multiple Myeloma and Non-Hodgkin Lymphoma. Biol Blood Marrow Transplant. 2017 Dec;23(12):2065-2069. doi: 10.1016/j.bbmt.2017.07.023. Epub 2017 Aug 7. PMID 28797783
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/20/2014 and closed to participant enrollment on 06/14/2016.
Groups:
- XM02 Filgrastim (Granix) and Plerixafor: XM02 Filgrastim (Granix) 10 mg/kg Days 1 through 4 (Days 5 through 8 may be required if target collection goal has not be met)
  Plerixafor 0.24 mg/kg Day 4 (Days 5 through 7 may be required if target collection goal has not be met)
  Apheresis on Day 5 (may need to be done on Days 6-8 if target collection goal has not been met)
- Filgrastim (Neupogen) and Plerixafor: Filgrastim (Neupogen) 10 mg/kg Days 1 through 4 (Days 5 through 8 may be required if target collection goal has not be met)
  Plerixafor 0.24 mg/kg Day 4 (Days 5 through 7 may be required if target collection goal has not be met)
  Apheresis on Day 5 (may need to be done on Days 6-8 if target collection goal has not been met)
Period: Overall Study
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Started | 49 | 51
Completed | 46 | 51
Not Completed | 3 | 0
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor | Total
Number analyzed (Participants) | 46 | 51 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.3) | 58.5 (9.0) | 60.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 38 | 47 | 85
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 51 | 97
Prior Therapies [Mean (Standard Deviation); unit: number of prior therapies] | 1.5 (0.8) | 1.4 (0.8) | 1.5 (0.8)
Diagnosis [Count of Participants; unit: Participants]
  Multiple myeloma | 43 | 43 | 86
  Non-Hodgkin's Lymphoma | 3 | 8 | 11
Prior Radiation [Count of Participants; unit: Participants] | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Mean Day 5 CD34+Cells/kg Yield Between the Two Arms
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: cells/kg
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 46 | 51
cells/kg | 11.6 (6.7) | 10.0 (6.8)

2. Secondary Outcome: Comparison of the Most Commonly Reported Adverse Events (Safety) Experienced by Participants Between the Two Arms
Description: -Adverse events will be assessed using CTCAE version 4.0
Time Frame: Up to 20 days after last apheresis (Day 25-Day 28)
Measure: Number; unit: participants
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 46 | 51
participants
  Bone pain | 19 | 22
  Thrombocytopenia | 18 | 20
  Anemia | 13 | 18
  Alkaline phosphatase increased | 10 | 12
  Nausea and/or vomiting | 10 | 10
  Leukocytosis | 8 | 10

3. Secondary Outcome: Comparison of the Time to Neutrophil Engraftment Between the Two Arms
Description: Time to neutrophil engraftment is measured by determining the first of 3 consecutive measurements of neutrophil count ≥ 500/µl following conditioning regimen-induced nadir. Patients who do not have neutrophil engraftment by Day 30 post-infusion of mobilized PBSC product will be considered a neutrophil engraftment failure.
Time Frame: Up to Day 30 post-infusion
Population: (2) participants in the XM02 Filgrastim (Granix) & Plerixafor arm did not receive ASCT and were not evaluable for this outcome measure. (1) participant in the Filgrastim (Neupogen) & Plerixafor arm did not receive ASCT and were not evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 44 | 50
days | 11 [11 to 12] | 11.5 [11 to 12]

4. Secondary Outcome: Comparison of the Time to Platelet Engraftment Between the Two Arms
Description: Time to platelet engraftment is measured by determining the first of 3 consecutive measurements of platelet count ≥ 50,000/µl without platelet transfusion support for 7 days. Patients who do not have platelet engraftment by Day 100 post-infusion of mobilized PBSC product will be considered a platelet engraftment failure.
Time Frame: Up to Day 100
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 44 | 50
days | 18 [16 to 21] | 17.5 [16 to 20]

5. Secondary Outcome: Comparison of the Readmission Rate Between the Two Arms
Description: Readmission rate is defined as the frequency at which patients are readmitted (after initial post-transplant discharge) following post-infusion of mobilized PBSC product for reasons other than progressive disease/relapse
Time Frame: Up to Day 100
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 44 | 50
Participants | 11 | 9

6. Secondary Outcome: Comparison of the Percentage of Patients Who Collect > 2.0x10^6 CD34+Cells/kg Following PBSC Mobilization Between the Two Arms
Time Frame: Up to Day 8 (total collection)
Measure: Number; unit: percentage of participants
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 46 | 51
percentage of participants | 100 | 100

7. Secondary Outcome: Comparison of the Percentage of Patients Who Collect > 5.0x10^6 CD34+Cells/kg Following PBSC Mobilization Between the Two Arms
Time Frame: Up to Day 8 (total collection)
Measure: Number; unit: percentage of participants
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 46 | 51
percentage of participants | 96 | 96

8. Secondary Outcome: Comparison of the Percentage of Patients Who Collect > 2.0x10^6 CD34+Cells/kg in One Apheresis Procedure Following PBSC Mobilization Between the Two Arms
Time Frame: Day 5
Measure: Number; unit: percentage of participants
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 46 | 51
percentage of participants | 98 | 90

9. Secondary Outcome: Comparison of the Percentage of Patients Who Collect > 5.0x10^6 CD34+Cells/kg in One Apheresis Procedure Following PBSC Mobilization Between the Two Arms
Time Frame: Day 5
Measure: Number; unit: percentage of participants
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Number analyzed (Participants) | 46 | 51
percentage of participants | 83 | 76

ADVERSE EVENTS:
Arm/Group | XM02 Filgrastim (Granix) and Plerixafor | Filgrastim (Neupogen) and Plerixafor
Serious Adverse Events (participants affected / at risk) | 2/46 | 3/51
Other Adverse Events (participants affected / at risk) | 45/46 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XM02 Filgrastim (Granix) and Plerixafor (N=46) | Filgrastim (Neupogen) and Plerixafor (N=51)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Edema - limbs (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Central line site cellulitis (Infections and infestations) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XM02 Filgrastim (Granix) and Plerixafor (N=46) | Filgrastim (Neupogen) and Plerixafor (N=51)
Anemia (Blood and lymphatic system disorders) | 13 | 18
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 8 | 10
Palpitations (Cardiac disorders) | 2 | 0
Scleral disorder (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Bloating (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 8
Oral dysesthesia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4
Chills (General disorders) | 1 | 5
Edema - limbs (General disorders) | 1 | 4
Fatigue (General disorders) | 0 | 3
Fever (General disorders) | 0 | 2
Injection site reaction (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 2
Pain (General disorders) | 1 | 0
Pain at biopsy site (General disorders) | 1 | 0
Pain at catheter site (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Rhinovirus positive culture (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Bleeding at catheter site (Injury, poisoning and procedural complications) | 5 | 4
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Discharge at catheter (Injury, poisoning and procedural complications) | 1 | 0
Drainage at catheter (Injury, poisoning and procedural complications) | 0 | 1
Erythema at catheter site (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Pain at catheter site (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 8 | 4
Alanine aminotransferase increased (Investigations) | 2 | 1
Alkaline phosphatase increased (Investigations) | 10 | 12
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 3 | 1
INR increased (Investigations) | 7 | 4
Lymphocyte count decreased (Investigations) | 18 | 21
Lymphocyte count increased (Investigations) | 15 | 10
Neutrophil count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 18 | 20
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 5 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 19 | 22
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hand cramping (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 3 | 4
Hypersomnia (Nervous system disorders) | 1 | 0
Movements involuntary (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Numbness of face (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 6 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 7 | 3
Confusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever blister (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes